CLINICAL TRIAL: NCT04536415
Title: Randomized, Open Label, Balanced, Two-Treatment, Two-Period, Two-Sequence, Single Dose, Crossover, Bioequivalence Study of Oseltamivir Phosphate 75 mg Capsule of Yangtze River Pharmaceutical (Group) Co., Ltd., China and TAMIFLU® (Oseltamivir Phosphate) Capsules 75 mg of Genentech, Inc., A Member of the Roche Group, 1 DNA Way, South San Francisco, CA 94080-4990 in Healthy, Adult, Human Subjects Under Fed Condition
Brief Title: Bioequivalence Study of Oseltamivir Phosphate and TAMIFLU Under Fed Condition in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Austarpharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20-VIN-0051
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oseltamivir Phosphate 75 mg capsules (Yangtze River) (Experimental): During the study session, healthy participants will be administered a single dose of Oseltamivir Phosphate capsules 75 mg of Yangtze River Pharmaceutical (Group) Co., Ltd., China under Fed condition.
  Interventions: Drug: Oseltamivir Phosphate 75 mg capsules
- Tamiflu capsules 75 mg (Genentech, Inc.) (Active Comparator): During the study session, healthy participants will be administered a single dose of Tamiflu capsules 75 mg of Genentech, Inc. under Fed condition.
  Interventions: Drug: Tamiflu capsules 75 mg

INTERVENTIONS:
Drug: Oseltamivir Phosphate 75 mg capsules — Capsules, 75 mg, single, oral dose
  Arms: Oseltamivir Phosphate 75 mg capsules (Yangtze River)
Drug: Tamiflu capsules 75 mg — Capsules, 75 mg, single, oral dose
  Arms: Tamiflu capsules 75 mg (Genentech, Inc.)

SUMMARY:
This study is to evaluate the bioequivalence of Oseltamivir Phosphate Capsules 75 mg versus TAMIFLU 75 mg capsules administered as 75 mg capsules in healthy volunteers under Fed condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' weight within normal range according to normal values for Body Mass Index (18.50 to 30.00 kg/m2) with minimum of 50 kg weight.
* Subjects with Hemoglobin level ≥ 11.5 G% at the time of screening.
* Subjects with normal health as determined by personal medical and medication history, clinical examination and laboratory examinations within the clinically acceptable normal range.
* Subjects having clinically acceptable 12-lead electrocardiogram (ECG).
* Subjects having clinically acceptable chest X-Ray (PA view).
* Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
* Subjects having negative alcohol breath test or urine alcohol test.
* Subjects willing to adhere to the protocol requirements and to provide written informed consent.
* For Male Subjects: Subjects willing to follow approved birth control methods (a double barrier method) for the duration of the study as judged by the investigator(s), such as (a double barrier method) condom with spermicide ,Condom with diaphragm , or abstinence, subjects should also not donate sperm during this time.
* Subjects having negative urine pregnancy test at screening and negative Serum β-hCG pregnancy test on admission day of period 01 (only for female subjects).
* For Female Subjects: Female of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as intrauterine device (IUD), or abstinence or double barrier contraception, i.e., condom + diaphragm, condom + spermicidal or foam; or Postmenopausal for at least 1 year, or if less than 1 year, then following acceptable contraceptive measures as mentioned above; Surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject).

Exclusion Criteria:

* Hypersensitivity to Oseltamivir or related class of drugs or any of its excipients or to heparin.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
* Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 30 days prior to dosing of period 01.
* Presence of significant alcoholism or drug abuse.
* History or presence of significant smoking (more than 10 cigarettes or beedis/day).
* History or presence of asthma, urticaria or other significant allergic reactions.
* History or presence of significant gastric and/or duodenal ulceration or gastrointestinal (GI) bleeding.
* History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
* History or presence of cancer or basal or squamous cell carcinoma.
* Difficulty with donating blood.
* Difficulty in swallowing solids like tablets or capsules.
* Use of any prescribed medication or OTC medication within 30 days prior to dosing in period 01.
* Major illness within past 3 months.
* Volunteer who have donated blood (1 unit) or participation in a drug research study within past 90 days prior to the first dose of the study drug.
* Consumption of xanthine-containing products, tobacco containing products or alcohol within 48 hours prior to dosing of period 01.
* Consumption of grapefruit or grapefruit juice containing products within 72 hours prior to dosing of period 01.
* Positive screening test result for any one or more: HIV, Hepatitis B and Hepatitis C.
* History or presence of significant easy bruising or bleeding.
* History or presence of significant recent trauma.
* Subjects who have been on an abnormal diet (for whatever reason) during the four weeks preceding the study.
* Female subjects who are currently breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Drug Concentration in Plasma After Single Dose Administration (Cmax) | 48 hours
  Maximum measured concentration over the time span specified
Area Under the Plasma Concentration Versus Time Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 48 hours
  The area under the concentration versus time curve, from time 0 to the last measurable concentration, where t = time of last measurable concentration, calculated using linear trapezoidal method
Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity After Single Dose (AUC) | 48 hours
  The area under the concentration versus time curve from time 0 to infinity AUC0-∞ = AUC0-t + Clast/Kel; where Clast is last measurable concentration, Kel is elimination rate constant.

CONTACTS AND LOCATIONS:
Overall Officials: Tejas Talati, MBBS, Principal Investigator — Veeda Clinical Research Pvt. Ltd
Locations (1):
- Austarpharma Llc, Edison, New Jersey, United States